CLINICAL TRIAL: NCT06654206
Title: Effects of a Strength Physical Exercise Program in Chronic Lymphocytic Leukemia Patients on Quality of Life, Mental Health, and Frailty.
Brief Title: Effects of a Strength Physical Exercise Program in Chronic Lymphocytic Leukemia Patients
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Salamanca (Other)
Collaborators: Colegio Profesional de Fisioterapeutas de Castilla y León (Unknown)
Responsible Party: Principal Investigator, CARLOS MARTIN SANCHEZ, PhD, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 21102024
Record Dates: First submitted 2024-10-21; First posted 2024-10-23 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Chronic Lymphocytic Leukemia; Exercise
Keywords: Exercise; Resistance; Chronic Lymphocytic Leukemia; Physiotherapy
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This is a double-blind, randomized controlled clinical trial with two parallel groups, in which patients diagnosed with Chronic Lymphocytic Leukemia (CLL) and undergoing active treatment will be recruited. Study participants will be assigned to one of two arms of the study: 1) Supervised Therapeutic Strength Exercise Intervention Group (GI); 2) Control Group without Supervised Exercise (GC). The study will last for 3 months. There will be 2 evaluation visits: one prior to the intervention (initial visit) and one at the end of the intervention (final visit). The intervention period will last for 8 weeks.
  The trial will be conducted following the CONSORT (Consolidated Standards of Reporting Trials) guidelines, and the current treatment protocol is described according to the SPIRIT (Standard Protocol Items: Recommendations for Interventional Trials) recommendations.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: In this research project, the evaluators will be blinded, as none of them will know which group the participants belong to. Due to the nature of the study, the participants cannot be blinded. Additionally, the statistical analysis will be performed by an independent statistician who will not be aware of the intervention group, and thus will also be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Therapeutic Strength Exercise Program): (Experimental): The therapeutic strength exercise program focused on strength exercises, although daily aerobic exercises were also included. The intervention group will participate in a supervised therapeutic strength exercise program twice a week, combined with a physical activity promotion program to be conducted at home three days a week. All supervised strength exercise sessions will be led by a physiotherapist in a physiotherapy clinic with appropriate space for the intervention.
  Interventions: Other: Exercise
- Control Group (CG), group without an exercise program (Active Comparator): Patients in the control group (CG) will only participate in the physical activity promotion program five days a week. This will be combined with walking for 60 minutes every day of the week.
  Interventions: Other: Home exercise

INTERVENTIONS:
Other: Exercise — Supervised strength exercise sessions: There will be two sessions per week, each lasting 50 minutes. Each session will consist of three distinct parts:
  Warm-up: 10 minutes of global strength and aerobic exercises at 6/10 on the Rating Perceived Exertion (RPE) scale.
  Strength training: 6 strength exercises targeting the major muscle groups, lasting 30 minutes. The initial load will be set at 70% of the estimated 1-RM (assessed in the first session and based on the individual patient). When the participant is able to complete 3 sets of 12 repetitions with the established weight in two consecutive sessions, the weight will be increased by 10%. The exercises will be performed in a circuit format with 30 seconds of rest between exercises and 90 seconds of rest between sets.
  Cool-down/stretching: 10 minutes of a combination of breathing exercises and stretching for the major muscle groups.
  Promotion of physical activity: Participants
  Arms: Intervention Group (Therapeutic Strength Exercise Program):
Other: Home exercise — Participants will complete three weekly home training sessions that will not coincide with supervised training days. Each session will last 20 minutes, they will complete two sets of five exercises, with one minute of work and one minute of rest.
  Arms: Control Group (CG), group without an exercise program

SUMMARY:
Chronic lymphocytic leukemia (CLL) is a hematological neoplasm that primarily affects older individuals and is the most common type of leukemia in adults in Western countries. CLL mainly affects older adults, with an average age at diagnosis of around 70 years, and there is a slightly higher risk in men compared to women. It is characterized by the proliferation of clonal B lymphocytes in peripheral blood, bone marrow, and lymphoid organs. Although CLL has a relatively slow progression in many cases, patients may experience chronic fatigue, muscle weakness, functional impairment, and psychological disorders, such as anxiety and depression, which significantly affect their quality of life.

In this context, it has been shown that physical exercise, especially strength training, can considerably improve physical and psychological conditions in oncology populations, such as those with breast cancer and colorectal cancer, as well as in older adults, where the benefits of resistance training are widely recognized. These benefits include increased muscle strength, reduced fatigue, improved functional abilities, psychological well-being, and overall quality of life. Furthermore, there is evidence that exercise can reduce systemic inflammatory markers, such as C-reactive protein (CRP), and improve lipid profiles by lowering total cholesterol and triglycerides, which is crucial for cancer patients at risk of cardiovascular diseases.

DETAILED DESCRIPTION:
Current research on the effects of physical exercise in patients with CLL is limited. While some studies suggest that cancer patients may benefit from physical exercise, most research has focused on other types of cancer, such as breast, lung, or colorectal cancer. In the case of patients with CLL, in addition to functional and psychological issues, they often experience chronic inflammation and alterations in lipid profiles, which can increase the risk of cardiovascular comorbidities.

Inflammatory markers, such as C-reactive protein (CRP) and pro-inflammatory cytokines (IL-6, TNF-α), are common in patients with CLL, and it has been suggested that modulating these markers through exercise may help control systemic inflammation. Strength training, in particular, could be beneficial for improving the inflammatory and lipid profiles in these patients, although this has not been thoroughly evaluated in this population.

Regarding mental health, studies have reported that patients with CLL experience high levels of anxiety and depression, which significantly deteriorate their quality of life. In other oncology populations, exercise has proven effective in reducing these symptoms and improving overall well-being. However, it has not been sufficiently studied whether these effects can be replicated in patients with CLL, representing a gap in the current literature.

Finally, the loss of muscle strength, a key indicator in the diagnosis of sarcopenia according to the diagnostic algorithm proposed by the European Working Group on Sarcopenia in Older People in 2019 (EWGSOP2), should be considered another common issue in patients with CLL, due to both the average age of the patients (70 years) and the disease itself or the side effects of treatment. Although it has been shown that physical exercise in general, and strength exercise in particular, can improve muscle strength and functional capacity in older adults and cancer patients, studies evaluating these effects in patients with CLL are lacking. Assessing how a strength training program can influence functional recovery and improve the quality of life of these patients is crucial for their clinical management.

ELIGIBILITY:
Inclusion Criteria

* Participants diagnosed with CLL or Small Lymphocytic Lymphoma (SLL) undergoing active treatment.
* Participants who have not engaged in regular physical activity in the past 8 weeks.
* Performance Status (ECOG) 0-1.
* Signed informed consent.

Exclusion Criteria

* The presence of any medical contraindications to physical exercise, such as severe musculoskeletal disorders, serious cardiovascular diseases, bone metastases, or other conditions as determined by a healthcare professional.
* Participants unable to complete the initial evaluation tests or who have difficulty performing basic exercises.
* Other circumstances, as determined by the researchers, that may interfere with the study's objectives or development.

Participants will be discontinued if they meet any of the following:

* Negative developments or progression of the tumor process.
* Severe adverse events related to exercise.
* Voluntary withdrawal from the intervention.
* New medical contraindications that prevent safe participation.
* Non-adherence to the intervention protocol that compromises study integrity.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Frailty | 8 weeks
  Frailty will be assessed using the Short Physical Performance Battery (SPPB) scale, which includes three components: a balance test, gait speed, and a chair stand test. The scale has a maximum score of 12 points, with higher scores reflecting better physical function.

SECONDARY OUTCOMES:
Quality of life | From enrollment to the end of the treatment, 8 weeks.
  Quality of life assessment: This will be conducted using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ). It is a general quality of life instrument for cancer patients. This questionnaire consists of 30 items, 24 of which are grouped into five functional scales (physical, role, emotional, cognitive, and social), three symptom scales (fatigue, pain, and nausea/vomiting), and one global health status scale. The remaining six items assess five symptoms (dyspnea, loss of appetite, insomnia, constipation, and diarrhea) and economic impact. A high score on the functional scale indicates greater functional capacity, while a high score on the symptom scale indicates greater distress.
Anxiety and depression | From enrollment to the end of the treatment, 8 weeks.
  Anxiety and depression assessment: These will be evaluated using the Hospital Anxiety and Depression Scale (HADS). The HADS is a reliable and valid questionnaire, consisting of seven questions (rated from 0 to 3) related to anxiety (subscale A) and another seven related to depression (subscale D), thus providing two separate scores.
Fatigue | From enrollment to the end of the treatment, 8 weeks.
  Fatigue assessment: This will be measured using the 13-item subscale of the Functional Assessment of Cancer Therapy-Fatigue (FACT-F). The FACT-F is a self-report questionnaire specifically designed to measure the degree of fatigue experienced by individuals with cancer and is the most widely used. It consists of 27 items in the general FACT section and an additional 13 items in the fatigue subscale, with scores ranging from 0 to 160. Higher scores on this scale indicate lower levels of fatigue.
Sleep quality | From enrollment to the end of the treatment, 8 weeks.
  Sleep quality assessment: The evaluation of insomnia will be conducted using the Athens Insomnia Scale. It consists of 8 items that assess sleep induction, awakenings during the night, early awakenings, duration, sleep quality, and daytime functioning. The response system is Likert-type, ranging from 0 (absence of the problem) to 3 (serious problem), and the overall score on the scale varies from 0 to 24 points.
Muscle strength | From enrollment to the end of the treatment, 8 weeks.
  The strength of both the lower and upper limbs will be assessed.The Jamar® dynamometer (J00105 Lafayette Instrument Company, USA), a hydraulic dynamometer considered the gold standard in the evaluation of grip strength, will be used. Both hands will be measured. The measurement will be performed following the Southampton Protocol. The patient will be seated in a chair with a backrest and the test will be explained to them. Three consecutive measurements will be taken on the same hand with a duration of 5 seconds per contraction and with an interval of 10 seconds between measurements. Encouraging commands will be given during the test to squeeze harder. The patient shall be seated in a chair with backrest, shoulder adducted and neutrally rotated, elbow flexed at 90°, forearm in neutral position and wrist in slight extension (0°-30°). The second Jamar® position shall be selected for all participants, with the exception of small hands which shall be placed in the first position.
Body composition | From enrollment to the end of the treatment, 8 weeks.
  Body composition assessment: The body mass index (BMI), appendicular lean mass (ALM), and estimated muscle mass will be calculated. This will be performed using electrical bioimpedance, which estimates muscle mass based on the electrical conductivity of the whole body. The TANITA BC-418 Body Composition Analyzer will be used.
Physical activity level | From enrollment to the end of the treatment, 8 weeks.
  Physical activity level assessment: This will be determined using the validated IPAQ-e questionnaire for older adults.
Physical performance | 8 weeks
  In addition to the SPPB, walking speed is assessed as a measure of physical performance associated with frailty using the four-meter walk test (4MWT). The patient starts walking one meter before the start line, where the stopwatch is activated, and is instructed to maintain his or her usual speed until four meters past the finish line. The test is performed three times, and the best value is recorded
Blood biomarker | From enrollment to the end of the treatment, 8 weeks.
  Blood biomarker assessment: A blood sample will be taken prior to the start of the exercise program and another within two weeks after its completion. Data from blood samples included in routine clinical practice will be collected to obtain lipid profile values. Additionally, a proteomic analysis of the samples will be conducted at the Cancer Research Center (Molecular and Cellular Biology of Cancer Institute - Laboratory 11 of Dr. Manuel Fuentes García).

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Martin Sanchez, PhD, Principal Investigator — University of Salamanca

IPD SHARING:
Plan to Share IPD: Yes
Further enquiries can be directed to the corresponding author. All the data collected in the study will be shared. Individual deidentified participant data are available. Additional and related documents such as study protocol or statistical analysis are available.
  The data will be available from April 2025 and for as long as necessary. The data will always be shared with the approval of the corresponding author analyzing the purpose which they are going to be used.
Supporting Information: SAP, ICF, CSR, Analytic Code
Time Frame: 2 years. From April 2025.
Access Criteria: Internet

REFERENCES:
- [Background] Brown JC, Spielmann G, Yang S, Compton SLE, Jones LW, Irwin ML, Ligibel JA, Meyerhardt JA. Effects of exercise or metformin on myokine concentrations in patients with breast and colorectal cancer: A phase II multi-centre factorial randomized trial. J Cachexia Sarcopenia Muscle. 2024 Aug;15(4):1520-1527. doi: 10.1002/jcsm.13509. Epub 2024 Jun 18. PMID 38887915
- [Derived] Sanchez-Gonzalez JL, Fernandez-Rodriguez EJ, Mendez-Sanchez R, Polo-Ferrero L, Puente-Gonzalez AS, de Ramon C, Marcos-Asensio S, Blazquez-Benito P, Navarro-Bailon A, Sanchez-Guijo F, Martin-Sanchez C. Effects of a strength physical exercise program in chronic lymphocytic leukemia patients on quality of life, mental health, and frailty: a randomized controlled trial study protocol. Front Sports Act Living. 2025 Mar 10;7:1534861. doi: 10.3389/fspor.2025.1534861. eCollection 2025. PMID 40129522